CLINICAL TRIAL: NCT03228654
Title: Electrosurgical Unipolar Vessel Sealing Versus Purohit Technique in Vaginal Hysterectomy . ( A Pilot Randomized Clinical Trial)
Brief Title: Electrosurgical Unipolar Vessel Sealing in Vaginal Hysterectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No available device in the hospital to complete study
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Abass, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Obs3514
Record Dates: First submitted 2017-07-21; First posted 2017-07-25 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Vaginal Hysterectomy
MeSH Terms: interventions — Hysterectomy, Vaginal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unipolar electrocautery (Experimental): vaginal hysterectomy using Unipolar electrocautery
  Interventions: Procedure: Unipolar Electrocautery sealing of vessels
- Purohit's technique (Active Comparator): Vaginal hysterectomy using Purohit's technique
  Interventions: Procedure: Purohit technique for vaginal hysterectomy

INTERVENTIONS:
Procedure: Unipolar Electrocautery sealing of vessels — 1. Vaginal walls are incised by monoplar current (40 W)
  2. A curved Bulldog Clamp is applied just 0.5 cm lateral to the uterine border along its attachements all through the pedicles. Then unipolar electrocautery (40 W) is applied to the pedicles along the lateral border of the uterus medial to the artery with maximum thickness 1 cm.
  3. uterine vessels are individually secured.
  4. Conventional volume reduction maneuvers are used as associated procedures in cases of large uteri to create the parauterine space to approach the lateral attachements.
  Other Names: Monopolar Electrocautery sealing of vessels
  Arms: Unipolar electrocautery
Procedure: Purohit technique for vaginal hysterectomy — using Bipolar electrosurgical sealing of vessels during vaginal hysterctomy
  Other Names: Bipolar electrosurgical sealing of vessels during vaginal hysterctomy
  Arms: Purohit's technique

SUMMARY:
Hysterectomy is one of the most common surgical procedures in gynecologic practice. Inspiteof the development of alternative treatments, the incidence of hysterectomy doesn't appear to be declining. Routes for hysterectomy include abdominal, vaginal, laparoscopic or combined approaches.Vaginal hysterectomy is the method of choice for removal of the uterus in patients with benign gynecological diseases. A Cochrane review of surgical approaches to hysterectomy for benign gynecological diseases concluded that, wee possible vaginal hysterectomy should be performed in preference to abdominal hysterectomy.

DETAILED DESCRIPTION:
A pilot prospective randomized clinical trial will be conducted at Ain shams University Maternity Hospital during the period from August 2016 to August 2018.

A sample size of 50 cases will be recruited from women presenting to the outpatient gynecologic clinic of Ain Shams University Maternity Hospital planned to undergo vaginal hysterectomy for benign cause. selected patients should be in age group from 40 to 70 years. Uterus size should be < 12 weeks with absence of significant scarring in the pelvis from previous surgeries. Endometriosis, Adnexal mass, malignancy, thinned out cervix should be excluded. After approval of the ethical committee , a detailed explanation of the procedure will e informed to the participant & her approval to be involved in the study, an informed written consent will be taken. After that, included patients will be randomized into 2 groups each one include 25 patients. First group includes women who will undergo vaginal hysterectomy using monopolar electrocautery. Second group includes women who will undergo vaginal hysterectomy using Purohit's technique. Principles of Purohit technique are 1. Vaginal walls are incised by monopolar current(30-50W).2.A right angle forceps is used o elevate, hook, stretch, spread and retract all the lateral attacements of uterus & vessels from their posterior aspects; tissues are coagulated using bipolar current (45 W) and divided between the prongs of forceps. 3. conventional volume reduction maneuvers are used as associated procedures in cases of large uteri to create the parauterine space for bipolar forceps and scissors.

Meanwhile the principles for vaginal hysterectomy using unipolar electrocautery are 1.Vaginal walls are incised by monopolar current(40 W) 2.A curved Bulldog clamp is applied just 0.5 cm lateral to uterine border along its attachements all through the pedicles. Then unipolar electrocautery (40 W) is applied to the pedicles along the lteral border of the uterus medial to the artery with maximum thickness 1 cm. 3. Uterine vessels are individually secured. 4. conventional volume reduction maneuvers are used as associated procedures in cases of large uteri to create the parauterine space for bipolar forceps and scissors.

ELIGIBILITY:
Inclusion Criteria:

* uterine size <12 weeks.
* presence of benign cause for the hysterectomy e.g. fibroid uterus, perimenopausal beeding not responding to medical treatment or complex endometrial hyperplasia without atypia.
* Absence of significant scarring in the pelvis from previous surgeries.

Exclusion Criteria:

* Suspected or known gynecological malignancy.
* uterine size >12 weeks.
* Endometriosis
* Presence of adnexal mass.
* cervix flushed with the vagina.
* presence of significant scarring in the pelvic area from previous surgery.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | 5 minutes after end if the procedure
  assessment of blood loss by assessing blood loss amount in suction bottle as well as soaked guzes and towels.

SECONDARY OUTCOMES:
operative time | 5 minutes after end of the procedure
  will be accounted from time of vaginal mucous membrane incision till closure of the vault.
postoperative pain | 6 hours postoperative
  pain scale will be used to assess pain
postoperative pain | 12 hours postoperative
  pain scale will be used to assess pain
postoperative pain | 24 hours postoperative
  pain scale will be used to assess pain
Hospital stay | 1 week after procedure
  number of days after the procedure the patient stay at the hospital

OTHER OUTCOMES:
postoperative complication | 1 week after procedure
  bleeding
postoperative complication | 1 week after procedure
  burns
postoperative complication | 1 week after procedure
  haemtoma
postoperative complication | 1 week after procedure
  urinary tract infections
postoperative complication | 1 week after procedure
  surgical site infection
postoperative complication | 1 week after procedure
  blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Tharwat, Ass. prof, Study Director — Ain Shams University; Amr H Yehia, Ass.prof, Study Chair — Ain Shams University; Alaa MA Karim El-din, ass. lect, Principal Investigator — Ain Shams University
Locations (1):
- Ahmed Abass, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR, Analytic Code